CLINICAL TRIAL: NCT01618786
Title: Randomized Controlled Trial of Compliant Flooring to Reduce Injuries Due to Falls in Older Adults in a Long-Term Care Facility
Brief Title: Flooring for Injury Prevention Trial
Acronym: FLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Stephen Robinovitch (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); AGE-WELL, Inc (Unknown); Fraser Health Authority (Unknown); Centre for Hip Health and Mobility (Unknown); New Vista Society Care Home (Unknown); Michael Smith Foundation for Health Research (Other); Canada Research Chair Program (Unknown); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Robinovitch, Professor, Department of Biomedical Physiology and Kinesiology, Simon Fraser University
Organization: Simon Fraser University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TIPS-001; TIR 103945 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2019-01

CONDITIONS: Accidental Falls; Bone Fracture; Traumatic Brain Injury; Head Injuries, Closed; Nursing Homes
Keywords: Falls; Fall injuries; Bone fracture; Hip fracture; Skull fracture; Wounds; Closed head injury; Traumatic brain injury; Concussion; Spinal cord injury; Trauma; Older adults; Long-term care; Compliant flooring; Safety floors; Balance; Injury biomechanics; Biomedical engineering; Environmental hazards; Environmental interventions; Fall prevention; Gerontology
MeSH Terms: conditions — Fractures, Bone; Brain Injuries, Traumatic; Head Injuries, Closed; Hip Fractures; Skull Fractures; Wounds and Injuries; Brain Concussion; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compliant Flooring (CF) (Experimental): Compliant flooring
  Interventions: Other: SmartCell flooring
- Control (CON) (Placebo Comparator): Non-compliant flooring
  Interventions: Other: Plywood flooring

INTERVENTIONS:
Other: SmartCell flooring — SmartCell (SATECH Inc., Chehalis, WA, USA) is a continuous rubber surface layer supported by an array of cylindrical rubber columns 14 mm in diameter, and spaced at 19 mm intervals. It has a surface hardness of 50 durometer. It has been reported to provide approximately 35% peak force attenuation during mechanical tests that simulate falls on the hip. It has also been reported to have minimal effect on balance and mobility of older women during activities of daily living. It will be covered with hospital-grade vinyl and will be inspected regularly for maintenance requirements.
  Arms: Compliant Flooring (CF)
Other: Plywood flooring — Plywood flooring covered with the same hospital-grade vinyl as the SmartCell flooring.
  Arms: Control (CON)

SUMMARY:
This study will evaluate the efficacy of novel compliant flooring in reducing injuries due to falls in a long-term care facility, determine the cost effectiveness of this intervention, and assess perceptions about compliant flooring among staff, residents, and families.

The investigators hypothesize that compliant flooring will (1) reduce the incidence of injuries due to falls in long-term care residents; (2) represent an overall cost-savings when material and implementation costs are considered relative to direct and indirect costs associated with injuries due to falls; and (3) be received positively by staff, residents, and their family members.

DETAILED DESCRIPTION:
Falls are the number one cause of unintentional injury among older adults in Canada, and are responsible for economic costs in excess of $1 billion CAD annually. In high-risk environments, such as long-term care (LTC) facilities, 60% of residents will experience at least one fall each year. Moreover, approximately 30% of falls in LTC residents result in injury, and 3 to 5% cause fractures.

A promising strategy for reducing the incidence of fall-related injuries in LTC facilities is to decrease the stiffness of the ground surface, and the subsequent force applied to the body parts at impact. Purpose-designed compliant flooring can reduce the force applied to the hip during a fall by up to 35 % (to allow a raw egg to be successfully bounced without cracking). Yet, few LTC facilities have flooring designed to reduce the impact of falls. This study will address this gap.

Resident rooms at a local LTC facility will be randomly assigned to installation of compliant flooring or control (non-compliant) flooring. Following installation, primary and secondary outcomes, including fall-related injuries and falls, will be monitored for 4 years and compared between resident rooms with and without compliant flooring. In addition, health resource utilization and their costs will be compared between resident rooms with and without compliant flooring. Perceptions about compliant flooring will be assessed among staff, residents, and their families.

ELIGIBILITY:
Inclusion Criteria (for rooms):

* Resident rooms across four units at New Vista Society Care Home, a long-term care facility in Burnaby, BC, Canada

Exclusion Criteria (for rooms):

* Resident rooms across four units at New Vista Society Care Home in which new flooring cannot be installed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Fall-related injuries | 4 years
  Moderate and serious injuries that result from falls in resident rooms. Assessed from incident and follow-up reports at participating long-term care facility.

SECONDARY OUTCOMES:
Falls | 4 years
  Falls in resident rooms. Assessed from incident reports at participating long-term care facility.
Fractures | 4 years
  Fractures in resident rooms. Assessed from incident and follow-up reports at participating long-term care facility.
Health resource utilization | 4 years
  Hospital transfers and admissions, emergency room visits, length of hospital stay, physician visits, physiotherapy and occupational therapy visits, nursing visits, diagnostic and lab procedures.
Musculoskeletal injuries | 4 years
  Work-related musculoskeletal injuries experienced by staff at participating long-term care facility.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn C Mackey, PhD, Principal Investigator — Simon Fraser University; Fabio Feldman, PhD, Principal Investigator — Fraser Health Authority; Andrew C Laing, PhD, Principal Investigator — University of Waterloo; Stephen N Robinovitch, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- New Vista Care Home, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lachance CC, Feldman F, Laing AC, Leung PM, Robinovitch SN, Mackey DC. Study protocol for the Flooring for Injury Prevention (FLIP) Study: a randomised controlled trial in long-term care. Inj Prev. 2016 Dec;22(6):453-460. doi: 10.1136/injuryprev-2016-042008. Epub 2016 Apr 4. PMID 27044272
- [Derived] Mackey DC, Lachance CC, Wang PT, Feldman F, Laing AC, Leung PM, Hu XJ, Robinovitch SN. The Flooring for Injury Prevention (FLIP) Study of compliant flooring for the prevention of fall-related injuries in long-term care: A randomized trial. PLoS Med. 2019 Jun 24;16(6):e1002843. doi: 10.1371/journal.pmed.1002843. eCollection 2019 Jun. PMID 31233541
- See also: Technology for Injury Prevention in Seniors (TIPS) — http://www.sfu.ca/tips